CLINICAL TRIAL: NCT00792337
Title: The Additive Anti-inflammatory Effect of Simvastatin in Combination With Inhaled Corticosteroids in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004(II)/51
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- simvastatin (Active Comparator): simvastatin in combination with budesonide
  Interventions: Drug: simvastatin
- B1-6-12 (Placebo Comparator): Budesonide in combination with B1-6-12
  Interventions: Drug: B1-6-12

INTERVENTIONS:
Drug: simvastatin — 10 mg per oral once daily for 8 weeks
  Other Names: zocor
  Arms: simvastatin
Drug: B1-6-12 — 1 table per day for 8 weeks
  Other Names: vitamin B1-6-12
  Arms: B1-6-12

SUMMARY:
We hypothesize that simvastatin in combination with ICS might have synergistic anti-inflammatory effects on airway inflammation in asthmatic patients

DETAILED DESCRIPTION:
To determine the additive effect of simvastatin on airway inflammation in ICS-treated patients with persistent asthma by measuring eosinophil counts in induced sputum

ELIGIBILITY:
Inclusion Criteria:

* He or she has FEV1 > 60% of predicted
* He or she requires less than 1000 mcg daily of beclomethasone or equivalent

Exclusion Criteria:

* He or she had previous history of renal disease or serum creatinine more than 2 mg/dL
* He or she had previous history of liver disease
* She is pregnant or during lactation
* He or she has already received statins or is allergic to statins or has developed myositis.
* He or she has an asthma exacerbation and requires treatment with oral corticosteroids during the 3 months prior to the commencement of study entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophil | 8 WEEKS

SECONDARY OUTCOMES:
FEV1 | 8 WEEKS
PC20 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong - Maneechotesuwan, MD, PhD, Principal Investigator — Siriraj Hospital
Locations (1):
- Kittipong Maneechotesuwan, Bangkoknoi, Bangkok, Thailand